CLINICAL TRIAL: NCT03934346
Title: Determination of Pre-Absorptive Dissociation of Zinc From a Zinc Amino Acid Complex in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-001
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Fractional Zinc Absorption
Keywords: zinc; absorption; kinetics; amino acid chelate

STUDY DESIGN:
Intervention Model Description: Nonlinear regression of fractional zinc absorption from 3 test diets using the Hill transport equation, and determination of an unknown amount of zinc based on fractional absorption from a single test diet. Order of the four test diets is randomized, with the constraint that the same oral zinc stable isotope tracer is not given on consecutive days.
Masking Description: Subjects are not informed of the amount of zinc in each test diet, or the order of the diets. The basic foods making up the test diets are identical in appearance and amount on each of the oral zinc stable isotope tracer days, so there is no way for the subject to distinguish any differences in the amount or form of zinc given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zinc transport kinetics (Other): Three different amounts of dietary zinc are used in the creation of a standard curve for determining zinc absorption kinetics: 4 mg, 7 mg, and 15 mg of zinc.
  Interventions: Other: Zinc amino acid complex

INTERVENTIONS:
Other: Zinc amino acid complex — Zinc in the form of a Zinc Amino Acid Complex (ZnAA) is provided with a test diet, and the amount of zinc that dissociates from the ZnAA and is thus absorbed via an ionic zinc transport pathway is determined based on the Hill transport kinetics for the respective subject.

SUMMARY:
Zinc may be absorbed from diet via zinc transporter mediated pathways, or, when coupled with amino acids, via amino acid transporter pathways. When zinc is coupled with amino acids in diet, it may dissociate from those amino acids in the acidic environment of the stomach prior to entering the small intestine. An experimentally-determined value for any pre-absorptive dissociation of zinc from a zinc amino acid complex (ZnAA) is necessary for the accurate compartmental modeling of zinc metabolism when provided as ZnAA compared with ionic zinc, which the investigators will perform in a future study. The current study will allow us to determine the dissociation of zinc from ZnAA, while serving as a pilot test of a novel technique to determine for the first time an individual's zinc transport kinetics.

DETAILED DESCRIPTION:
An experimentally-determined value for any pre-absorptive dissociation of zinc from ZnAA is necessary for the accurate compartmental modeling of zinc metabolism when provided as ZnAA compared with zinc chloride, which the investigators will perform in a future study.

The current study will allow us to determine the pre-absorptive dissociation of zinc from ZnAA, while serving as a pilot test of a novel technique to determine for the first time an individual's zinc transport kinetics. Since zinc absorption kinetics follow a saturable process, the zinc transport maximum (Tr_max) and transport rate (K_Tr) can be determined by fitting Hill transport equation to measurements of absorbed zinc at 3 or more levels of zinc intake (mg zinc/d):

Total Absorbed Zinc (TAZ) = (Zinc Intake * Tr_max) / (Zinc Intake + K_Tr)

Although population data have been used to estimate zinc transport kinetics (Tran, et al. AJCN 2004), Tr_max and K_tr have never been determined in individual subjects. The investigators plan to determine the fractional zinc absorption (FZA) from multiple levels of dietary zinc in rapid succession (Chung, et al. AJCN 2004) and, therefore, estimate an individual's transport maximum and rate, Tr_max and K_Tr. Once Tr_max and K_Tr are known, the FZA can be used to determine an unknown zinc intake from zinc chloride and any zinc dissociated from the ZnAA complex using the following equation:

Zinc Intake = (Tr_max / FZA) - K_Tr

Since zinc that dissociates from the ZnAA complex will compete for absorption with the inorganic zinc stable isotopic oral tracer (70-zinc chloride), reducing the amount of that tracer absorbed, the investigators can therefore determine the total zinc intake (the sum of the known zinc in the controlled study diet and the unknown quantity of zinc dissociated from ZnAA pre-absorption) based on the transport kinetics (FZA, Tr_max and KTr).

In other words, for the meal with added ZnAA, the zinc intake is the sum of the zinc in the test meal (3.6 mg zinc and 0.4 mg 70-Zn tracer) and the zinc that dissociates from the ZnAA complex pre-absorption. Since the intact ZnAA (i.e. that zinc that does not dissociate pre-absorption from the ZnAA complex) is absorbed by a different transport mechanism (Sauer, et al. Biometals 2017), it does not compete with the stable isotope tracer for absorption via zinc cation transporters and is, therefore, not part of the "zinc intake" for the purpose of these calculations.

If the hypothesized 20% dissociation is correct (i.e. 3 mg zinc dissociated from an initial 15 mg ZnAA), the total amount of ionic zinc will be 7 mg (the 3.6 mg base diet, 0.4 mg zinc stable isotope tracer, and 3 mg dissociated zinc), and the FZA will therefore be the same as that from a 7 mg test diet (the 3.6 mg base diet, 0.4 mg zinc tracer, and 3 mg zinc as zinc chloride).

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men
* Body mass index between 18 and 30 kg/m2
* Willing to eat only the foods provided by the study for a 2 week period

Exclusion Criteria:

* Those reporting any chronic or acute diseases, food allergies, smoking or alcohol abuse
* Use of illicit drugs; regular consumption of medications, micronutrient supplements, or both
* Vegetarians, or those unable to eat meat, are also excluded since the foods for the study contain meat
* Unable to refrain from taking medications during the study period

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Zinc Transport Curve | 2 weeks
  The saturable zinc transport curve determined by fitting the zinc absorption data to the Hill transport equation
Dissociated Amino Acid Zinc | 2 weeks
  Amount of zinc dissociated from the ZnAA prior to absorption

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hall, Ph.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Children's Hospital and Research Center Oakland, Oakland, California, United States

REFERENCES:
- [Background] Chung CS, Stookey J, Dare D, Welch R, Nguyen TQ, Roehl R, Peerson JM, King JC, Brown KH. Current dietary zinc intake has a greater effect on fractional zinc absorption than does longer term zinc consumption in healthy adult men. Am J Clin Nutr. 2008 May;87(5):1224-9. doi: 10.1093/ajcn/87.5.1224. PMID 18469243
- [Background] Tran CD, Miller LV, Krebs NF, Lei S, Hambidge KM. Zinc absorption as a function of the dose of zinc sulfate in aqueous solution. Am J Clin Nutr. 2004 Dec;80(6):1570-3. doi: 10.1093/ajcn/80.6.1570. PMID 15585770
- [Background] Sauer AK, Pfaender S, Hagmeyer S, Tarana L, Mattes AK, Briel F, Kury S, Boeckers TM, Grabrucker AM. Characterization of zinc amino acid complexes for zinc delivery in vitro using Caco-2 cells and enterocytes from hiPSC. Biometals. 2017 Oct;30(5):643-661. doi: 10.1007/s10534-017-0033-y. Epub 2017 Jul 17. PMID 28717982